CLINICAL TRIAL: NCT06975527
Title: Milk Production and Body Weight Response to Suggested Protocol in Obese Lactating Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Elshafei, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003736
Record Dates: First submitted 2025-05-06; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding guidelines group (Active Comparator): The participants will receive breastfeeding guidelines for 6 weeks
  Interventions: Other: Breastfeeding guidelines
- Aerobic exercise and breastfeeding guidelines (Experimental): The participants will receive aerobic exercises for 40 minutes, 3 times per week in addition to breastfeeding guidelines for 6 weeks.
  Interventions: Other: Breastfeeding guidelines; Other: Aerobic exercise

INTERVENTIONS:
Other: Breastfeeding guidelines — All participants will be instructed by the following guidelines:
  * Hold the breast so the nipple brushes the center of the infant's lips and wait for the infant to open the mouth.
  * Infant's mouth should be opened wide, as with a yawn and should cover the entire areola, or a large amount of the areola.
  * Both breasts are used in each feeding, usually 10 to 15 minutes on the first side, followed by burping before beginning the second side.
  * Break suction by placing finger in the corner of infant's mouth and quickly remove breast.
  * Apply breast massage before breastfeeding.
  * The neonate is nursed shortly after birth and approximately every 2 to 3 hours thereafter for a total of 8 to 12 feedings a day.
  * Lactating women needs about 8 to 10 glasses of fluids per day while breastfeeding.
  * Caffeine consumption should be limited to 2 cups of coffee, tea or cola per day.
  * Lactating mother should consume a healthy diet which is varied, balanced, and natural.
Other: Aerobic exercise — The participants will be engaged in a supervised moderate aerobic exercise in the form of walking on a treadmill for 40 minutes/ day, 3 days/ week, for 6 weeks beginning 6:8 weeks postpartum. Each exercise session will be divided into 3 phases. The warm-up phase begins with walking at low speed (within resting heart rate) on a treadmill for 5 minutes. The active phase continues for 30 minutes at a moderate intensity of 60 to 70% of maximal heart rate (HRmax). Gradual increase and adjustment of speed will be applied for each woman according to her prescribed intensity based on HRmax. HRmax is calculated by subtracting the age from 220. The program will be terminated with 5 minutes cool-down phase, during which the treadmill speed will be gradually decreased until the heart rate resumes its resting level.
  Arms: Aerobic exercise and breastfeeding guidelines

SUMMARY:
This study will investigate the milk production and body weight response of both mother and the newborn to aerobic exercise in obese lactating women.

DETAILED DESCRIPTION:
Breastfeeding is a normal method of providing nutrition to young infant by breast milk. Breastfeeding is equally important and beneficial for not only infant but also for the mother.

Women with high BMI have delays in establishing lactation after giving birth. In addition, overweight and obesity increase the risk of early cessation of breastfeeding.

Aerobic exercises have positive effects on breastfeeding frequency and body weight of neonate and can increase blood flow to the chest which is effective in lactation performance.

So, this study will help to evaluate the efficacy of aerobic exercise in addition to guidelines for breastfeeding, nutrition and fluid intake on milk production, baby and mother weight.

ELIGIBILITY:
Inclusion Criteria:

* Multiparous obese mothers having number of parity ranges from two to four times.
* Lactating mothers within 2nd month after delivery.
* All of them diagnosed by gynecologist as having insufficient lactation
* Age will range from 25-35 years old.
* Body mass index: 30-40 Kg/m².

Exclusion Criteria:

* Lactating women suffering from postpartum hemorrhage
* Poor mammary development
* Cardio respiratory disease
* Diabetes mellitus
* Breast cancer
* Getting pregnant again during breast feeding period
* Mental disorders
* Previous surgeries in the chest, breast or the surrounding area
* Anemia
* Having twins or causes that hindering normal breast feeding as (mastitis, retracted, cracked, inflamed or inverted nipple)

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of the degree of improvement in the flow of milk | 6 weeks
  Each lactating mother in both groups will have a visual analogue scale (VAS) form containing a straight line its ends are defined as the extreme limits of milk flow. The mother will select the suitable description of her milk flow before and after the end of the treatment procedures. The scale ranged from 0-4. 0 means no milk flow. 4 means extreme milk flow.
Serum prolactin level | 6 weeks
  ELISA Kit will be used for quantitative determination of the human prolactin concentration in serum. it will be measured for all lactating women before and after the treatment. Normal prolactin level is ranged from 100:110 ng/ml.
Weight of the baby | 6 weeks
  The baby will be weighed in kilograms at the beginning and after the end of treatment period by placing the baby over the baby weight scale wearing only the underwear and the baby diapers are removed.
Weight of the mother | 6 weeks
  The lactating mother will be weighed in kilograms by the weight scale while wearing a thin layer of clothes and with bare feet to assess and compare her weight before and after the end of the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Afaf Botla, Professor, Study Director — Cairo University; Dalia Kamel, Professor, Study Chair — Cairo University
Locations (1):
- Mai mohamed mohamed Elshafei, Beheira, Egypt